CLINICAL TRIAL: NCT04091555
Title: Evaluation of the Impact of the HL Natural, Inc. Tension Relief Product on the Reduction of Symptoms in Adults Who Suffer From Mild to Moderate Tension Headaches
Brief Title: Evaluation of the Impact of the HL Natural, Inc. Tension Relief Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawthorne Effect Inc. (Other)
Collaborators: HLNatural, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00037556
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Tension; Headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients who suffer from symptoms of tension headaches (Other): Patients will begin taking the capsules at the onset of headache symptoms.
  Interventions: Dietary Supplement: HLNatural Tension

INTERVENTIONS:
Dietary Supplement: HLNatural Tension — Understand the impact of the supplement on Tension Headaches

SUMMARY:
The primary hypothesis of the present study is that supplementation with the Tension Relief test product will reduce the severity of symptoms of a tension headache.

DETAILED DESCRIPTION:
Patients will begin taking the capsules at the onset of headache symptoms. Onset is defined as the point in time the participant feels that it is necessary to take the test product for relief of symptoms. When the participant decides to take the test product, they will report symptoms in the headache diary prior to taking the product and rate their symptoms on a 10-point Mankoski scale. After consuming the product, the participant will complete a Mankoski scale at 15 minutes, 30 minutes and 1 hour after taking the product. If needed the participant will be allowed to take alternative medication (alternative treatment) after an hour after taking the product. If alternative medication is taken, the participant will record this in their headache diary.

ELIGIBILITY:
Inclusion Criteria:

Adult candidates who are in overall good health and who suffer from mild to moderate tension headaches.

Participants will be deemed to be in good health if they do not report any of the existing medical conditions asked about in the screening questionnaire.

Exclusion Criteria:

* Those who have been diagnosed with migraine headaches.
* Those who score between 36-49 or 60-78 on screening questionnaire.
* Is < 18 years of age
* Those who have been diagnosed with fibromyalgia.
* Women that are pregnant or breastfeeding.
* Alcohol consumption more than 7 drinks per week or more than 3 drinks per occasion.
* Routine recreational drug use such as marijuana.
* Chronic renal disease
* Chronic liver disease
* Allergy to any of the following: Aspirin or any other product including Salicylates, Boswellia, Feverfew, Skullcap, White Willow Bark, Rice Hull, or Vegetable Cellulose.
* Unable to swallow pills.
* Unwilling to try test product for relief of pain and tension headache symptoms.
* Participants who are currently taking any anticoagulation medications daily. (Aspirin, Warfarin, Heparin etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2020-08-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
The Evaluation of the Impact of HLNatural Tension Relief Product for Adults who Suffer from Mild to Moderate Tension Headaches | After taking the test product, the participant will complete a Mankoski pain scale at 15 minutes after the start of the event, 30 minutes after the start of the event, and 1 hour after the start of the event.
  Those subjects who meet the inclusion/exclusion criteria will be invited to be part of the study. The subject will sign consent and complete the required surgery and questionnaires before taking the test product. • At the onset of the headache, the participant will start a Headache Diary and complete a 10-point Mankoski pain scale. • After completing the surveys, the participant will take test product. The participant will take 2 capsules with 6-8 oz. of water per headache episode. With a max of 6 pills per day.

SECONDARY OUTCOMES:
Understanding If HLNatural impacts the Intensity of Tension Headaches. Headaches.another intervention | Stubjects will be evaluated for up to 60 days or 3 episodes of a headache
  A diary will be kept of the intensity and need for other intervention during each episode.
Outcome of all Adverse Events while consuming HLNatural Suppliement | All adverse events will be captured throughout the 60 days or after 3 episodes of headaches or until the subject exits the trial.
  Throughout the study the subject will capture any adverse events that have occurred. All events will recorded in the subject's diary.
Outcome of Subjects Natural Behavior During the Clinical Trial | 10-point Mankoski Scale and Headache Diary will be at the start of the headache, 15 minutes after start of the event, 30 minutes after start of event and 60 minutes after the start of the event. The activity will be repeated for up to 3 events.
  Before the test product is taken the subject will complete a screening, demographic and baseline survey. At the end of the survey the researchers will use what is in the literature to help establish normal behavior. Upon completion of the study the participant will complete an exit study. The surveys and questionnaires will be used to establish normal behavior of the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Soyona Rafatjah, MD, Principal Investigator — Hawthorne Effect Inc.
Locations (1):
- Hawthorne Effect, Inc., Lafayette, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. 15 Pain Scales (And How to Find The Best Pain Scale For You). (2018, January 05). Retrieved from https://paindoctor.com/pain-scales/
- [Background] Beer AM, Wegener T. Willow bark extract (Salicis cortex) for gonarthrosis and coxarthrosis--results of a cohort study with a control group. Phytomedicine. 2008 Nov;15(11):907-13. doi: 10.1016/j.phymed.2008.07.010. Epub 2008 Sep 23. PMID 18815018
- [Background] Cady RK, Goldstein J, Nett R, Mitchell R, Beach ME, Browning R. A double-blind placebo-controlled pilot study of sublingual feverfew and ginger (LipiGesic M) in the treatment of migraine. Headache. 2011 Jul-Aug;51(7):1078-86. doi: 10.1111/j.1526-4610.2011.01910.x. Epub 2011 Jun 1. PMID 21631494
- [Background] Ertsey C, Magyar M, Gyure T, Balogh E, Bozsik G. [Tension type headache and its treatment possibilities]. Ideggyogy Sz. 2019 Jan 30;72(1-2):13-21. doi: 10.18071/isz.72.0013. Hungarian. PMID 30785242
- [Background] 5. Friedman, L. M., Furberg, C., DeMets, D. L., Reboussin, D., & Granger, C. B. (2015). Fundamentals of clinical trials. Cham: Springer.
- [Background] Kimmatkar N, Thawani V, Hingorani L, Khiyani R. Efficacy and tolerability of Boswellia serrata extract in treatment of osteoarthritis of knee--a randomized double blind placebo controlled trial. Phytomedicine. 2003 Jan;10(1):3-7. doi: 10.1078/094471103321648593. PMID 12622457
- [Background] 7. Kubala, J., MS, RD. (2019, April 30). Skullcap: Benefits, Side Effects, and Dosage. Retrieved from https://www.healthline.com/nutrition/skullcap
- [Background] Riva A, Allegrini P, Franceschi F, Togni S, Giacomelli L, Eggenhoffner R. A novel boswellic acids delivery form (Casperome(R)) in the management of musculoskeletal disorders: a review. Eur Rev Med Pharmacol Sci. 2017 Nov;21(22):5258-5263. doi: 10.26355/eurrev_201711_13849. PMID 29228442
- [Background] Pareek A, Suthar M, Rathore GS, Bansal V. Feverfew (Tanacetum parthenium L.): A systematic review. Pharmacogn Rev. 2011 Jan;5(9):103-10. doi: 10.4103/0973-7847.79105. PMID 22096324
- [Background] Prabhavathi K, Chandra US, Soanker R, Rani PU. A randomized, double blind, placebo controlled, cross over study to evaluate the analgesic activity of Boswellia serrata in healthy volunteers using mechanical pain model. Indian J Pharmacol. 2014 Sep-Oct;46(5):475-9. doi: 10.4103/0253-7613.140570. PMID 25298573
- [Background] 11. Taylor, F. R. (2018, November 17). Tension-type headache in adults: Pathophysiology, clinical features, and diagnosis. Retrieved from https://www.uptodate.com/contents/tension-type-headache-in-adults-pathophysiology-clinical-features-and-diagnosis
- [Background] 12. The R Project for Statistical Computing. (n.d.). Retrieved from https://www.R-project.org/.
- [Background] 13. Vitamin C. (2017, October 18). Retrieved from https://www.mayoclinic.org/drugs-supplements-vitamin-c/art-20363932
- [Background] 14. Willow Bark Uses, Benefits & Dosage. (n.d.). Retrieved from https://www.drugs.com/npp/willow-bark.html
- [Background] 15. Wu, B. (n.d.). Magnesium glycinate: Uses, benefits, and side effects (A. Carter PharmD, Ed.). Retrieved from https://www.medicalnewstoday.com/articles/315372.php
- [Background] Schwartz BS, Stewart WF, Simon D, Lipton RB. Epidemiology of tension-type headache. JAMA. 1998 Feb 4;279(5):381-3. doi: 10.1001/jama.279.5.381. PMID 9459472
- [Background] Jensen R, Stovner LJ. Epidemiology and comorbidity of headache. Lancet Neurol. 2008 Apr;7(4):354-61. doi: 10.1016/S1474-4422(08)70062-0. PMID 18339350
- [Background] Douglas ME, Randleman ML, DeLane AM, Palmer GA. Determining pain scale preference in a veteran population experiencing chronic pain. Pain Manag Nurs. 2014 Sep;15(3):625-31. doi: 10.1016/j.pmn.2013.06.003. Epub 2014 Feb 14. PMID 24530196
- [Background] Majeed M, Majeed S, Narayanan NK, Nagabhushanam K. A pilot, randomized, double-blind, placebo-controlled trial to assess the safety and efficacy of a novel Boswellia serrata extract in the management of osteoarthritis of the knee. Phytother Res. 2019 May;33(5):1457-1468. doi: 10.1002/ptr.6338. Epub 2019 Mar 6. PMID 30838706
- [Background] Nahrstedt A, Schmidt M, Jaggi R, Metz J, Khayyal MT. Willow bark extract: the contribution of polyphenols to the overall effect. Wien Med Wochenschr. 2007;157(13-14):348-51. doi: 10.1007/s10354-007-0437-3. PMID 17704985
- [Background] Fiebich BL, Chrubasik S. Effects of an ethanolic salix extract on the release of selected inflammatory mediators in vitro. Phytomedicine. 2004 Feb;11(2-3):135-8. doi: 10.1078/0944-7113-00338. PMID 15070163
- [Background] Chrubasik S, Eisenberg E, Balan E, Weinberger T, Luzzati R, Conradt C. Treatment of low back pain exacerbations with willow bark extract: a randomized double-blind study. Am J Med. 2000 Jul;109(1):9-14. doi: 10.1016/s0002-9343(00)00442-3. PMID 10936472
- [Background] Gagnier JJ, Oltean H, van Tulder MW, Berman BM, Bombardier C, Robbins CB. Herbal Medicine for Low Back Pain: A Cochrane Review. Spine (Phila Pa 1976). 2016 Jan;41(2):116-33. doi: 10.1097/BRS.0000000000001310. PMID 26630428
- [Background] Oltean H, Robbins C, van Tulder MW, Berman BM, Bombardier C, Gagnier JJ. Herbal medicine for low-back pain. Cochrane Database Syst Rev. 2014 Dec 23;2014(12):CD004504. doi: 10.1002/14651858.CD004504.pub4. PMID 25536022
- [Background] 25. Skullcap monograph. Engles, G. Herbalgram. The American Botanical Council. Issue 83, pg 1-2
- [Background] Brock C, Whitehouse J, Tewfik I, Towell T. American Skullcap (Scutellaria lateriflora): a randomised, double-blind placebo-controlled crossover study of its effects on mood in healthy volunteers. Phytother Res. 2014 May;28(5):692-8. doi: 10.1002/ptr.5044. Epub 2013 Jul 22. PMID 23878109
- [Background] Johnson ES, Kadam NP, Hylands DM, Hylands PJ. Efficacy of feverfew as prophylactic treatment of migraine. Br Med J (Clin Res Ed). 1985 Aug 31;291(6495):569-73. doi: 10.1136/bmj.291.6495.569. PMID 3929876
- [Background] Murphy JJ, Heptinstall S, Mitchell JR. Randomised double-blind placebo-controlled trial of feverfew in migraine prevention. Lancet. 1988 Jul 23;2(8604):189-92. doi: 10.1016/s0140-6736(88)92289-1. PMID 2899663
- [Background] 29. Palevitch D, Earon G, Carasso R. Feverfew (tanacetum parthenium) as a prophylactic treatment for migraine- a double-blind, placebo-controlled study. Phytotherapy Res 1997;11:508-11.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/55/NCT04091555/Prot_SAP_ICF_000.pdf